CLINICAL TRIAL: NCT04595669
Title: Personalised Dietary Advice for Highly Motivated Consumers at Risk of Metabolic Syndrome - a Pilot Study
Brief Title: Personalised Advice for the Prevention of Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: TNO (Other); Philips Healthcare (Industry); Friesland Campina (Unknown); Albert Heijn (Unknown); Menzis (Unknown); Smart with food (Unknown); Vital-10 (Unknown); Dutch Spices (Unknown)
Responsible Party: Principal Investigator, Diederik Esser, Researcher, PhD, Wageningen University and Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NL61382.028.17
Record Dates: First submitted 2020-10-15; First posted 2020-10-20 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Metabolic Syndrome, Protection Against
Keywords: personalised dietary advice; metabolic syndrome; dietary behaviour
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalised advice (Experimental)
  Interventions: Behavioral: Personalised advise

INTERVENTIONS:
Behavioral: Personalised advise — personalised dietary advice in combination with feedback on dietary behaviour and health status (i.e. waist circumference, blood pressure, cholesterol, glucose and triglycerides)

SUMMARY:
Rationale: Improving dietary behaviours in view of optimising risk factors of metabolic syndrome requires behaviour change strategies. Tailored dietary advice, i.e. recommendations offered as a guide to action, can support behaviour change. In the current study we aim to learn how to better help consumers in their daily life to make lifestyle choices that better match their personal health target than their usual choices by providing personalised advice and feedback. In this study we target consumers at risk of metabolic syndrome (MetS) that are highly motivated to change their dietary behaviour in view of improving health.

Objective: The primary objective is to investigate the potential of personalised dietary advice and feedback for initiating and maintaining dietary changes by consumers at risk of MetS. In addition we want to evaluate understanding, applicability and personal benefit of personalised dietary advice and feedback by the target population to be able to further optimize the personalisation in future studies. The secondary objective is to explore potential effects of personalised dietary advice and feedback on subjective health and metabolic health parameters.

Study design: The study follows a one group pre-test post-test design with a duration of 16 weeks after the first advice is provided to the participants.

Study population: In total 40 adult men and women at risk of metabolic syndrome will be recruited from the consumer databases of Wageningen Food & Biobased Research. Consumers are eligible for study participation when they are highly motivated to change dietary behaviour, willing to use technology, willing to share food purchase data as registered on a customer card of the supermarket, and in possession of a smart-phone.

Intervention: The intervention consists of personalised dietary advice and feedback on actual behaviour and health status that will be provided to study participants at set time points throughout the study period. The content of the advice will be generated partly automated based on dietary intake and parameters of metabolic health using knowledge rules that are developed for this study. During a consultation with the dietician, the advice is then translated in a dietary behaviour change strategy by taking into account individual preferences through motivational interviewing.

Main study parameters/endpoints: Primary outcomes of the study are the adequacy of intake of fruits, vegetables, whole grain products, dairy, fish, fats & oils, red meat, processed meat, and sweetened beverages & fruit juices as estimated by the online tool Eetscore. Furthermore consumer experiences and individual benefits of the provided personalised dietary advice are monitored on a weekly basis throughout the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Having given written informed consent
* Aged 40 years or over
* At risk of metabolic syndrome
* Motivated to change behaviour
* Willing to use technology (digital platforms, activity tracker, digital questionnaires, apps)
* Customer of supermarket Albert Heijn (at least 1x per week) and in possession of customer card
* Willing to share food purchase data as registered with the Bonuskaart with the investigators
* In possession of I-phone or mobile phone with android system

Exclusion Criteria:

* Use of medication known for its effects on blood glucose, cholesterol or insulin
* Suffering from diabetes
* Familial hypercholesterolemia
* Following a specific diet
* Having an alcohol consumption > 28 units/week for males and > 21 units (drinks)/week for females
* Does not accept that the general practitioner will be informed about participation of the study
* Having holidays planned for a period of more than two weeks during the intervention period

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Dietary quality at baseline | Baseline (week 0)
  Dietary quality was assessed by an online version of the Dutch Healthy Diet Index (DHDI) ('Eetscore', Division of Human Nutrition, Wageningen University). The DHDI evaluates adherence to the Dutch dietary guidelines per food category (score 1-10) and a total score (score 8-80).
Dietary quality halfway | halfway (week 8)
  Dietary quality was assessed by an online version of the Dutch Healthy Diet Index (DHDI) ('Eetscore', Division of Human Nutrition, Wageningen University). The DHDI evaluates adherence to the Dutch dietary guidelines per food category (score 1-10) and a total score (score 8-80).
Dietary quality at study end | study end (week 16)
  Dietary quality was assessed by an online version of the Dutch Healthy Diet Index (DHDI) ('Eetscore', Division of Human Nutrition, Wageningen University). The DHDI evaluates adherence to the Dutch dietary guidelines per food category (score 1-10) and a total score (score 8-80).
Consumer experiences | study end (week 16)
  Questionnaire to evaluate experiences with personalized advice and feedback
Changes in Self perceived health during study period | Baseline (week 0) and study end (week 16)
  questionnaire to evaluate 1-self-perceived health status, 2-healthiness of the diet and 3-satisfaction with actual diet. Items All items were evaluated on a 7-point scale. For items 1 and 2, the scale ranged from 1=very unhealthy up to 7=very healthy. For item 3, the scale ranged from 1=very unsatisfied up to 7=very satisfied

SECONDARY OUTCOMES:
Waist circumference | Baseline (week 0), halfway (week 8) and study end (week 16)
  in cm
Body weight | Baseline (week 0), halfway (week 8) and study end (week 16)
  measured on a calibrated weighing scale to the nearest 0.1 kg
Blood pressure | Baseline (week 0), halfway (week 8) and study end (week 16)
  in mmHg, measured in finger prick blood by research nurse with the Medisana upper-arm blood pressure monitor
Lipid profile (HDL and LDL cholesterol, triglycerides) | Baseline (week 0), halfway (week 8) and study end (week 16)
  measured in finger prick blood by research nurse by the Mission Cholesterol 3-1 device
Glucose | Baseline (week 0), halfway (week 8) and study end (week 16)
  measured in finger prick blood by research nurse by the Meditouch 2 device
C-peptide | Baseline (week 0), halfway (week 8) and study end (week 16)
  assessed in dried blood spots by high performance liquid chromatography with ultraviolet detection and liquid chromatography mass spectrometry
Carotenoids in blood | Baseline (week 0), halfway (week 8) and study end (week 16)
  assessed in dried blood spots by high performance liquid chromatography with ultraviolet detection and liquid chromatography mass spectrometry

CONTACTS AND LOCATIONS:
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] van der Haar S, Hoevenaars FPM, van den Brink WJ, van den Broek T, Timmer M, Boorsma A, Doets EL. Exploring the Potential of Personalized Dietary Advice for Health Improvement in Motivated Individuals With Premetabolic Syndrome: Pretest-Posttest Study. JMIR Form Res. 2021 Jun 24;5(6):e25043. doi: 10.2196/25043. PMID 34185002